CLINICAL TRIAL: NCT02508064
Title: A Two-Part Study to Evaluate the Bioavailability of BMS-626529 Administered as Prodrug BMS-663068 From Prototype Low-Dose Extended-Release Tablets (Part 1) and Prototype Multi-Particulate Formulations (Part 2) Relative to the 600 mg Extended Release Tablet in Healthy Subjects
Brief Title: Bioavailability of BMS-626529 in Healthy Subjects From Prototype Low Dose Extended Release Formulations (Part 1) and Prototype Extended Release Multi-particulate Formulations (Part 2) of BMS-663068 Relative to 600 mg Extended Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 206288; AI438-054 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part 1 (Experimental): BMS-663068 1 × 600 mg extended-release (ER) tablet formulation
  Interventions: Drug: BMS-663068
- Part 1: Prototype 1 (Experimental): BMS-663068 600 mg ER low-dose tablet formulation (Prototype 1)
  Interventions: Drug: BMS-663068
- Part 1: Prototype 2 (Experimental): BMS-663068 600 mg ER low-dose tablet formulation (Prototype 2)
  Interventions: Drug: BMS-663068
- Part 1: Prototype 3 (Experimental): BMS-663068 600 mg ER low-dose tablet formulation (Prototype 3)
  Interventions: Drug: BMS-663068
- Part 1: Prototype 4 (Experimental): BMS-663068 600 mg ER low-dose tablet formulation (Prototype 4)
  Interventions: Drug: BMS-663068
- Part 1: Prototype 5 (Experimental): BMS-663068 600 mg ER low-dose tablet formulation (Prototype 5)
  Interventions: Drug: BMS-663068
- Part 2 (Experimental): BMS-663068 1 × 600 mg ER tablet formulation
  Interventions: Drug: BMS-663068
- Part 2: Prototype 1 (Experimental): BMS-663068 600 mg ER prototype multi-particulate formulation (Prototype 1)
  Interventions: Drug: BMS-663068
- Part 2: Prototype 2 (Experimental): BMS-663068 600 mg ER prototype multi-particulate formulation (Prototype 2)
  Interventions: Drug: BMS-663068
- Part 2: Prototype 3 (Experimental): BMS-663068 600 mg ER prototype multi-particulate formulation (Prototype 3)
  Interventions: Drug: BMS-663068
- Part 2: Prototype 4 (Experimental): BMS-663068 600 mg ER prototype multi-particulate formulation (Prototype 4)
  Interventions: Drug: BMS-663068

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068

SUMMARY:
This 2-part study will determine the bioavailability of BMS-626529 in healthy subjects from prototype low dose extended release formulations (Part 1) of BMS-663068 and prototype extended release multi-particulate formulations (Part 2) of BMS-663068 relative to 600 mg extended release tablet of BMS-663068.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and females, 18 to 50 years of age, inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical and surgical history, PE findings, vital sign measurements, 12-lead ECG measurements, physical measurements, and clinical laboratory test results
* Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (performed for all females; minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study drug

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Evidence of organ dysfunction or any clinically significant deviation from normal in PE, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population
* Any of the following on 12-lead ECG prior to study drug administration, confirmed by repeat:

  i) PR ≥ 210 msec ii) QRS ≥ 120 msec iii) QT ≥ 500 msec and iv) QTcF ≥ 450 msec
* Exposure to any investigational drug or placebo within 12 weeks of study drug administration
* Positive blood screen for hepatitis C antibody (HCV Ab), hepatitis B surface antigen (HBsAg), or HIV-1 and HIV-2 antibody

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of BMS-626529 | Day 1 to Day 4 of each period
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) of BMS-626529 | Day 1 to Day 4 of each period
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-626529 | Day 1 to Day 4 of each period

SECONDARY OUTCOMES:
Safety of BMS-663068 will be measured by incidence of Adverse events (AEs), Serious adverse events (SAEs), and AEs leading to discontinuation;, and results of clinical laboratory tests, vital signs, 12-lead ECGs, and Physical examination (PE) | Day 1 to Day 4 of each period; for SAEs up to 30 days post discontinuation of dosing
Tolerability of BMS-663068 will be measured by incidence of AEs, SAEs, and AEs leading to discontinuation; and results of clinical laboratory tests, vital signs and 12-lead ECGs | Day 1 to Day 4 of each period; for SAEs up to 30 days post discontinuation of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom